CLINICAL TRIAL: NCT02144792
Title: Development and Clinical Application of [11C]Verapamil-PET, a Surrogate Marker on P-glycoprotein Expression
Brief Title: Development and Clinical Application of [11C]Verapamil-PET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Kun Lee, Seoul National University Hospital, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0720130520
Record Dates: First submitted 2014-04-22; First posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (healthy persons) (Active Comparator): Normal controls take a [11C] -verapamil PET scan. While P-gp inhibitor (Cyclosporin A, 2.5mg/kg/hr during 2hours, intravenous) is infused, PET scans were done using [11C] -verapamil, a substrate of P-gp.
  Interventions: Drug: [11C] -verapamil PET
- Patients with drug-resistant epilesy (Active Comparator): Patients with drug-resistant epilepsy take a [11C] -verapamil PET scan. While P-gp inhibitor (Cyclosporin A, 2.5mg/kg/hr during 2hours, intravenous) is infused, PET scans were done using [11C] -verapamil, a substrate of P-gp.
  Interventions: Drug: [11C] -verapamil PET
- Patients with drug-sensitive epilepsy (Active Comparator): Patients with drug-sensitive epilepsy take a [11C] -verapamil PET scan. While P-gp inhibitor (Cyclosporin A, 2.5mg/kg/hr during 2hours, intravenous) is infused, PET scans were done using [11C] -verapamil, a substrate of P-gp.
  Interventions: Drug: [11C] -verapamil PET

INTERVENTIONS:
Drug: [11C] -verapamil PET — While P-gp inhibitor (Cyclosporin A, 2.5mg/kg/hr during 2hours, intravenous) is infused, PET scans were done using [11C] -verapamil, a substrate of P-gp.
  Other Names: VPM PET

SUMMARY:
The major hypothesis explaining drug resistance is overexpression of p-glycoprotein at the target lesion. Based on several studies, p-glycoprotein (P-gp) has an important role in neurologic diseases, especially in drug resistant epilepsy. But there is no surrogate marker that can quantify the expression of P-gp because of the difficulty in measuring substances in the neurologic system and the lack of clinical trials. Here, the investigators use a novel non-invasive [11C] -verapamil Brain PET and SPAM analytic method as a surrogate marker for quantifying the expression of p-glycoprotein.

DETAILED DESCRIPTION:
A pilot study on healthy volunteers and a case-control study on patients with drug resistant epilepsy and drug sensitive epilepsy is performed. The investigators compare the whole brain SUV in each group (normal control, drug resistant epilepsy, drug sensitive epilepsy) and the asymmetry by the standardized uptake value(SUV) of ipsilateral areas and contralateral areas.

[11C] -verapamil PET will be used as a surrogate marker of P-gp expression in patients with epilepsy, and will be an important prognostic factor of individualized drug therapy. Also, it can be used as a biomarker in checking of the drug efficacy of novel medications. Furthermore, by localizing epileptogenic zones for patients, [11C] -verapamil PET could contribute in improving the prognosis of surgical treatment in drug resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy controls ( age range 20-45 years)
* Patient age (> 15), diagnose as epilepsy

Exclusion Criteria:

* Subjects who take medicines that affect on the function of p-glycoproteins
* Pregnancy or subject who feed the breast milk
* Subjects who had severe renal disease or liver disease
* Subjects who need treated by immunosuppressant or take immunosuppressant

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Measured Asymmetric index[(SUV in Right regions - SUV in Left regions)/(SUV in Right regions+ SUV in left regions)] in all three groups | first visit day
  Comparing with Asymmetry index in each groups

SECONDARY OUTCOMES:
Number of patients with side effect of cyclosporine and [11C]-verapamil PET | During and after the drug injection, During and after the PET Scan [first visit day]

CONTACTS AND LOCATIONS:
Overall Officials: Sang Kun Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea